CLINICAL TRIAL: NCT03498222
Title: Phase I Study in Patients With Tumours Requiring Arginine to Assess ADI-PEG 20 With Atezolizumab, Pemetrexed and Carboplatin (ADIAtezoPemCarbo) (iTRAP Study)
Brief Title: Study in Patients With Tumours Requiring Arginine to Assess ADI-PEG 20 With Atezolizumab, Pemetrexed and Carboplatin
Acronym: iTRAP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funder and IMP manufacturer withdrew support
Sponsor: Queen Mary University of London (Other)
Collaborators: Polaris Group (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 012375QM
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Pemetrexed; Carboplatin; ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dose Level -1 (Experimental): Atezolizumab 1200mg Pemetrexed 500mg/m2 Carboplatin AUC5 ADI PEG20 9mg/m2
  Interventions: Drug: Atezolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: ADI PEG20
- Dose Level 1 (Experimental): Atezolizumab 1200mg Pemetrexed 500mg/m2 Carboplatin AUC5 ADI PEG20 18mg/m2
  Interventions: Drug: Atezolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: ADI PEG20
- Dose Level 2 (Experimental): Atezolizumab 1200mg Pemetrexed 500mg/m2 Carboplatin AUC5 ADI PEG20 36mg/m2
  Interventions: Drug: Atezolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: ADI PEG20

INTERVENTIONS:
Drug: Atezolizumab — Administered at a fixed dose of 1200 mg (equivalent to an average body weight-based dose of 15mg/kg) by intravenous (IV) infusion every 3 weeks (21 days).
  Other Names: Tecentriq
Drug: Pemetrexed — Administered at a fixed dose of 500mg/m2 by IV infusion every 3 weeks.
  Other Names: Alimta
Drug: Carboplatin — Administered at a fixed dose of AUC5 by IV infusion every 3 weeks.
Drug: ADI PEG20 — Administered by intramuscular (IM) injection to patients once weekly.

SUMMARY:
iTRAP is an open-label, multi-centre, dose escalation study of ADI PEG20 in combination with atezolizumab, pemetrexed and carboplatin in patients with advanced non-squamous non-small cell lung carcinoma (NSCLC) - stage IIIB/IV.

DETAILED DESCRIPTION:
iTRAP is an open-label, multi-centre, dose escalation study of ADI PEG20 in combination with atezolizumab, pemetrexed and carboplatin in patients with advanced non-squamous NSCLC (stage IIIB/IV). Patients will initially receive 4 cycles of ADI PEG20 in combination with atezolizumab, pemetrexed and carboplatin unless there is documented disease progression or unacceptable toxicities. On completion of 4 cycles and in the absence of disease progression requiring other therapeutic interventions, patients may receive additional cycles of ADI PEG20 and/or atezolizumab and/or pemetrexed for up to a maximum of 2 years at the discretion of the treating physician.

Dose escalation will occur using a 3 + 3 design. The trial will start at dose level 1, which represents 100% of the recommended dose of carboplatin (AUC5) and pemetrexed (500mg/m2) when given as a combination, 100% of the atezolizumab recommended dose (1200mg) and 50% of the recommended single agent dose of ADI PEG20 (18mg/m2). ADI PEG20 doses will be increased according to pre-planned dose escalations.

If the maximum tolerated dose (MTD) is reached with the first 6 patients, up to an additional 6 patients will be enrolled at the MTD. The MTD is defined as the dose level below that at which 2/3 or ≥3/6 patients experience a dose limiting toxicity (DLT).

The maximum administered dose (MAD) may also equal the MTD if dose escalation is stopped before two DLTs are observed at a given dose level due to the expectation that higher dose levels would be too toxic to administer to patients or the maximum planned dose level has been achieved.

The MTD will be determined following review of all the relevant toxicity data by the Safety Review Committee (SRC).

If dose level 1 equals the MAD then dose level -1 may be investigated with a 50% reduction in ADI PEG20 (9mg/m2) along with atezolizumab 1200mg, carboplatin AUC5, and pemetrexed 500mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to study entry.
* Age ≥ 18 years.
* Histologically proven advanced non-squamous NSCLC (stage IIIB/IV) not treated with chemotherapy or immunotherapy - immunotherapy for uveal melanoma and prior (neo)adjuvant chemotherapy is permitted. Patients with EGFR mutant or ALK positive NSCLC must have had an EGFR tyrosine kinase inhibitor (TKI) or ALK inhibitor and progressed or been shown to be intolerant of therapy prior to enrolling in this trial.
* ASS1 deficiency defined as ≤50% ASS expression on tissue specimen by immunohistochemistry (IHC) (cytospin samples are acceptable) - assessed centrally. For patients previously treated with (neo)adjuvant chemotherapy, this specimen may have been obtained before that chemotherapy.
* Measurable disease as assessed by RECIST 1.1 i.e. at least one lesion, not previously irradiated, that can be measured accurately at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements OR lytic or mixed (lytic + sclerotic) bone lesions in the absence of measurable disease as defined above; NOTE: patients with sclerotic / osteoblastic bone lesions only in the absence of measurable disease are not eligible)
* ECOG performance status of 0 - 1
* Fully recovered from any prior surgery and no major surgery within 4 weeks of initiating study treatment. Surgery for placement of vascular access devices is acceptable.
* Female patients of childbearing potential and their partners (if male) and male patients with female partners of childbearing potential and their partners must agree to use a highly effective form of contraception for the duration of the study and until 35 days after the final dose of ADI-PEG 20 or 180 days after the final dose of atezolizumab, pemetrexed or carboplatin, whichever is later.
* Negative serum or urine pregnancy test for female patients of childbearing potential within 14 days prior to cycle 1 day 1.
* Adequate normal organ, marrow and coagulation function within 28 days prior to cycle 1 day 1
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits and examinations including follow up.

Exclusion Criteria:

* Radiotherapy (including for palliative reasons) or targeted therapywithin four weeks before study treatment.
* History of autoimmune disease
* Ongoing toxic manifestations of previous treatments.
* Symptomatic brain or spinal cord metastases (patients must be stable for > 3 months post radiotherapy or surgery).
* Major thoracic or abdominal surgery from which the patient has not yet recovered.
* Serious infection requiring treatment with intravenous antibiotics at the time of study entrance, or an infection requiring intravenous therapy within 7 days prior to the first dose of study treatment.
* Known to be serologically positive for human immunodeficiency virus (HIV).
* Known active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Uncontrolled serious intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, and social situations that would limit compliance with study requirements.
* Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within 8 weeks of study treatment.
* Ongoing therapeutic anticoagulation (prophylactic dose low molecular weight heparin is acceptable).
* Concurrent treatment with other experimental drugs or participation in another interventional clinical study with therapeutic intent within 28 days from cycle 1 day 1. Participation in an observational or biomarker study would be acceptable, with prior Sponsor approval.
* Malignancies other than NSCLC within 5 years prior to study entry, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome.
* Prior treatment with cluster of differentiation 137 (CD137) agonists, anti-cytotoxic-T-lymphocyte-associated antigen 4 (anti-CTLA4), anti-programmed death-1 (anti-PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanised antibodies or fusion proteins.
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation.
* Prior allogeneic stem cell or solid organ transplantation.
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computerised tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis.
* Receipt of a live, attenuated vaccine within 4 weeks prior to cycle 1 day 1 or anticipation that a live, attenuated vaccine will be required during atezolizumab treatment or within 5 months after the last dose of atezolizumab.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to cycle 1 day 1.
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities | First 21 days of treatment
  Protocol defined haematological events attributed as possibly, probably or definitely related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szlosarek, Study Chair — Queen Mary University of London